CLINICAL TRIAL: NCT02125331
Title: Measurement of NonInvasive Blood Pressure With DINAMAP SuperSTAT and Datex-Ohmeda With Intra-arterial Blood Pressure in Neonates Through Adults and Special Populations
Brief Title: Measurement of NonInvasive Blood Pressure in Neonates Through Adults and Special Populations
Acronym: MISSION
Status: Terminated | Type: Observational
Why Stopped: Data collection requirment complete
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 123.04-2013-GES-0008
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Blood Pressure
Keywords: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PDM-SuperSTAT: PDM-SuperSTAT Arm (minimum of 55 evaluable patients): GE DINAMAP® SuperSTAT algorithm delivered by the PDM acquisition module connected to the CARESCAPE Monitor B650
  Interventions: Procedure: Device: Blood pressure monitoring with GE Healthcare CARESCAPE B650 Patient Monitor-Patient Side Module (PSM) or Patient Data Module (PDM)
- PSM-Datex-Ohmeda: PSM-Datex-Ohmeda Arm (minimum of 45 evaluable patients): Datex-Ohmeda delivered by the PSM acquisition module connected to the CARESCAPE Monitor B650
  Interventions: Procedure: Device: Blood pressure monitoring with GE Healthcare CARESCAPE B650 Patient Monitor-Patient Side Module (PSM) or Patient Data Module (PDM)

INTERVENTIONS:
Procedure: Device: Blood pressure monitoring with GE Healthcare CARESCAPE B650 Patient Monitor-Patient Side Module (PSM) or Patient Data Module (PDM) — 3-15 Non-Invasive Blood Pressure readings on the CARESCAPE B650 Patient Monitor equipped with PSM-Datex-Ohmeda and PDM-SuperSTAT NIBP measurement devices during non-emergent heart catheterization
  Other Names: GE Healthcare CARESCAPE B650 Patient Monitor; Patient Side Module with Datex-Ohmeda software algorithm (PSM); Patient Data Module with SuperSTAT software algorithm (PDM)

SUMMARY:
This study is required to demonstrate that the non-invasive blood pressure (NIBP) measurement algorithms on two commercially available multifunction hemodynamic acquisition modules, the Patient Data Module (PDM) equipped with the DINAMAP® SUPERSTAT algorithm ("PDM-SUPERSTAT") and the Patient Side Module (PSM) equipped with Datex-Ohmeda GE algorithm ("PSM-Datex-Ohmeda"), provide accurate NIBP measurements in accordance with the guidelines provided by the most recent International Organization for Standardization (ISO) 81060-2:2013.

Notably, the new ISO 81060-2:2013 supersedes the previous 2009 version of this standard, and this study is being conducted in accordance with the most recent applicable standards.

This study will assess neonate, infant, children, pediatric, adolescent, and adult patients as well as adults with chronic atrial fibrillation in a population that requires non-emergent heart catheterization.

This is a study conducted to satisfy both standards for two NIBP devices and, as such, does not require a statistical hypothesis.

DETAILED DESCRIPTION:
This study is required to demonstrate that the non-invasive blood pressure (NIBP) measurement algorithms on two commercially available multifunction hemodynamic acquisition modules, the Patient Data Module (PDM) equipped with the DINAMAP® SUPERSTAT algorithm ("PDM-SUPERSTAT") and the Patient Side Module (PSM) equipped with Datex-Ohmeda GE algorithm ("PSM-Datex-Ohmeda"), provide accurate NIBP measurements in accordance with the guidelines provided by the most recent International Organization for Standardization (ISO) 81060-2:2013.

Notably, the new ISO 81060-2:2013 supersedes the previous 2009 version of this standard, and this study is being conducted in accordance with the most recent applicable standards.

This study will assess neonate, infant, children, pediatric, adolescent, and adult patients as well as adults with chronic atrial fibrillation in a population that requires non-emergent heart catheterization.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects will be included that:

1. Are aged >29 days requiring clinically indicated non-emergent heart catheterization OR aged ≤29 days with placed or scheduled placement of an indwelling femoral, radial, or umbilical arterial monitoring line;
2. Have an upper limb (right OR left side) that fits a cuff size of the device (circumference ranging 3 cm to 40 cm) OR have a thigh (right OR left side) that fits a cuff size of the device (circumference ranging 38 to 50 cm);
3. Are expected to be able to provide blood pressure measurements using both IBP and NIBP;
4. Are able and willing to provide written informed consent or have a legally authorized representative willing to provide written informed consent with assent from minor patients, as required by IRB policy.

EXCLUSION CRITERIA

Subjects will be excluded that:

1. Have previously participated in this study (no subject may participate more than once).
2. Exhibit signs or symptoms or have a current diagnosis of peripheral vascular disease in either upper AND/OR lower limbs;
3. Have current, uncontrolled circulatory shock;
4. Exhibit injuries, deformities, intravenous lines, or other abnormalities that, in the opinion of the investigator, may prevent proper cuff application or functioning;
5. For women of child-bearing potential, are currently pregnant, suspected to be pregnant, or are currently lactating;
6. Have any condition that could interfere with the subjects ability to tolerate the procedure, including having a maximum of 4 fast flushes (adult, adolescent, or pediatric patients aged >29 days) or 1 fast flush (neonates aged <29 days);
7. If aged greater than 29 days but less than 12 years of age, have previously had any clinical or research procedure requiring general anesthesia in the last 3 month period;
8. If aged greater than 29 days but less than 12 years of age, are expected to require more than three (3) total hours of continuous general anesthesia for the scheduled procedure (including clinically necessary anesthesia and anticipated 25 minute extension for study purposes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include neonates with indwelling femoral, radial, or umbilical arterial monitoring lines and infant, pediatric, adolescent, and adult subjects requiring non-emergent surgery involving aortic catheterization (including chronic atrial fibrillation patients among adults and adolescents).
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Marks, MD, MBA, Principal Investigator — Medical College of Wisconsin
Locations (4):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Wheaton Franciscan Healthcare - St. Joseph's, Milwaukee, Wisconsin
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- NH Narayana Multispecialty Hospital, Unit of Narayana Health Mazumdar Shaw Medical Center, Bangalore, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PDM-SuperSTAT | PSM-Datex-Ohmeda
Started | 58 | 25
Completed | 53 | 25
Not Completed | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — technical problem | 2 | 0
Not completed — screen failure | 2 | 0

BASELINE CHARACTERISTICS:
Population: Total of subjects enrolled and assigned to PDM-SuperSTAT arm or PSM-Datex-Ohmeda arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | PDM-SuperSTAT | PSM-Datex-Ohmeda | Total
Number analyzed (Participants) | 58 | 25 | 83
Age, Customized [Count of Participants; unit: Participants]
  Subjects >= 3 years | 34 | 19 | 53
  Subjects < 3 years | 24 | 6 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 13 | 38
  Male | 33 | 12 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Subjects with Chronic Atrial Fibrillation [Count of Participants; unit: Participants] | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate NIBP Measurements as Confirmed by IBP Measurements
Description: Comparison of the following measurements: non-invasive blood pressure to invasive blood pressure. This is done with a beat to beat comparison. Each pulse from the analyzed time interval (non-invasive blood pressure determination) provides a systolic, MAP and diastolic value and that is compared to the waveform collected at the same timepoint for the invasive BP (measurement). Criteria is defined in ANSI/AAMI/ISO 81060-2 NIBP Standard. Mean & SD of the IBP derived from the IBP wave recordings during a NIBP determination will be calculated; and the range of reference IBP will be determined as mean ±1 standard deviation (SD) of the IBPs. The same method will be used for both systolic and diastolic blood pressures. Data may be excluded for analysis when the range of invasive systolic BP is wider than 20 mmHg or when the range of invasive diastolic BP is wider than 12 mmHg, as such that analysis is performed in accordance with ISO 81060-2:2013.
Time Frame: 60 minutes
Population: The PDM-SuperSTAT arm was analyzed according to the ISO 81060-2:2013(E) standard. As the PSM-Datex-Ohmeda was prematurely terminated, PASS/FAIL criteria were unable to be determined.
Measure: Count of Participants; unit: Participants
Groups:
- PDM-SuperSTAT: PDM-SuperSTAT Arm (minimum of 55 evaluable patients): GE DINAMAP® SuperSTAT algorithm delivered by the PDM acquisition module connected to the CARESCAPE Monitor B650
  The result of the analysis of mean blood pressure measurement errors shows the PDM-SuperSTAT arm population groups ≥ 3 years old and < 3 years old passed the acceptance criteria. However, the Chronic AFib subgroup population of ≥ 3- years old did not meet the subject enrollment because of the challenging population; but as a group, the NIBP determinations for the PDM-SuperSTAT arm for both population group of ≥ 3 years old and < 3 years old showed the study conformed to ISO 81060-2:2013(E) standards.
- PSM-Datex-Ohmeda: PSM-Datex-Ohmeda Arm (minimum of 45 evaluable patients): Datex-Ohmeda delivered by the PSM acquisition module connected to the CARESCAPE Monitor B650
  For the PSM-Datex-Ohmeda arm population group ≥ 3 years old and < 3 years old that was prematurely terminated as a result of the business decision that the data was no longer needed to satisfy the business requirements, as a whole, did not meet the ISO 81060-2:2013(E) standards; therefore, PASS/FAIL criteria were unable to be determined.
Arm/Group | PDM-SuperSTAT | PSM-Datex-Ohmeda
Number analyzed (Participants) | 53 | 25
Participants | 40 | 19

ADVERSE EVENTS:
Time Frame: The duration over which adverse events were monitored/assessed was 2 hours.
Arm/Group | PDM-SuperSTAT | PSM-Datex-Ohmeda
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/25
Other Adverse Events (participants affected / at risk) | 3/58 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDM-SuperSTAT (N=58) | PSM-Datex-Ohmeda (N=25)
Cuff irritation (Injury, poisoning and procedural complications) | 2 (2) | NA
Heart Block (Surgical and medical procedures) | 1 (1) | NA — Complete heart block secondary to catheter placement not study procedure.

LIMITATIONS AND CAVEATS:
Terminated prematurely due to the challenging recruitment of Atrial Fibrillation Patients- PDM arm and PSM arm was prematurely terminated as a result of the business decision that the data was no longer needed to satisfy the business requirements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications using study data, in full or in part, will be subject to approval by the Sponsor prior to submission. The Investigator and Sponsor agree to act in good faith to consider the interests of each party in publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT02125331/Prot_SAP_000.pdf